CLINICAL TRIAL: NCT01156922
Title: B-lymphocyte Depletion Using the Monoclonal Anti-CD20 Antibody Rituximab in Severely Affected Chronic Fatigue Syndrome Patients. An Open Label Phase II Study With Rituximab Induction and Maintenance Treatment for Patients in WHO Performance Status III-IV
Brief Title: B-cell Depletion Using the Monoclonal Anti-CD20 Antibody Rituximab in Very Severe Chronic Fatigue Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties in logistics handling the very severe patients (travel, hospital stay, follow-up)
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010/1321
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Chronic Fatigue Syndrome; Myalgic Encephalomyelitis
Keywords: Chronic fatigue syndrome; CFS; Myalgic encephalomyelitis; Rituximab; B-cell depletion
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab (Experimental): Rituximab induction two infusions (500 mg/m2, max 1000 mg) two weeks apart, followed by maintenance Rituximab infusions (500 mg/m2, max 1000 mg) after 3, 6, 10 and 15 months.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Two infusions of Rituximab 500 mg/m2 (max 1000 mg) given two weeks apart, followed by maintenance Rituximab infusions 500 mg/m2 (max 1000 mg) at 3, 6, 10, and 15 months.
  For up to 5 patients in the study, standard plasma exchange (one plasma volume, up to 5 treatments, during 1-2 weeks) will be performed 2-3 weeks prior to start of Rituximab therapy.
  Amendment: for patients with gradual improvement in CFS/ME symptoms after 12 months follow-up, but not having reached a clear response, up to 6 additional Rituximab infusions (500 mg/m2, max 1000 mg) may be given during the following 12 months period.

SUMMARY:
Based on pilot patient observations, and experience from the prior study KTS-1-2008, the investigators anticipate that severely affected chronic fatigue syndrome patients may benefit from B-cell depletion therapy using Rituximab induction with maintenance treatment.

The hypothesis is that at least a subset of chronic fatigue syndrome (CFS) patients have an activated immune system involving B-lymphocytes, and that prolonged B-cell depletion may alleviate symptoms.

An approved amendment (April 15th 2011): the study will be extended with up to 5 patients. For up to 5 patients in the study, standard plasma exchange may be performed 2-3 weeks prior to start of B-lymphocyte depletion using Rituximab (as in the protocol).

Approved amendment (December 2011): for patients with gradual improvement in CFS/ME symptoms after 12 months follow-up, but not having reached a clear response, up to 6 additional Rituximab infusions (500 mg/m2, max 1000 mg) may be given during the following 12 months period.

ELIGIBILITY:
Inclusion Criteria:

* patients severely affected by chronic fatigue syndrome, in WHO performance status III or IV.
* age 18-66 years
* informed consent

Exclusion Criteria:

* patients with fatigue, not fulfilling criteria for CFS
* pregnancy or lactation
* previous malignant disease except basal cell carcinoma of skin and cervical carcinoma in situ
* previous major immunological disease, except autoimmune diseases such as diabetes mellitus or thyroiditis
* endogenous depression
* lack of ability to comply by the protocol
* multi-allergy with risk of serious drug reaction
* reduced renal function (creatinin > 1.5 x upper normal limit [UNL])
* reduced liver function (bilirubin or transaminases > 1.5 x UNL)
* HIV positivity
* evidence of clinically significant infection

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Symptom alleviation, as compared to baseline, measured by standardized self-reports and quality of life schemes | Major response of at least six weeks duration, independent on when occuring, during the follow-up period
  The primary endpoint is defined as major response of the CFS symptoms, of at least six weeks duration, independent on when during 36 months follow-up the response period(s) occurs. Single such response periods, and the sum of these, are recorded.

SECONDARY OUTCOMES:
Symptom alleviation, as compared to baseline, measured by standardized self-reports and quality of life schemes. | At 3, 6, 10, 15, 20, 24, 30, 36 months after intervention
  The secondary outcome measures are effect on the CFS symptoms, by evaluation at 3, 6, 10, 15, 20, 24, 30, and 36 months after first intervention (i.e. first Rituximab infusion)

CONTACTS AND LOCATIONS:
Overall Officials: Olav Mella, PhD, MD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Department of Oncology and Medical Physics, Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Background] Fluge O, Mella O. Clinical impact of B-cell depletion with the anti-CD20 antibody rituximab in chronic fatigue syndrome: a preliminary case series. BMC Neurol. 2009 Jul 1;9:28. doi: 10.1186/1471-2377-9-28. PMID 19566965
- [Result] Fluge O, Risa K, Lunde S, Alme K, Rekeland IG, Sapkota D, Kristoffersen EK, Sorland K, Bruland O, Dahl O, Mella O. B-Lymphocyte Depletion in Myalgic Encephalopathy/ Chronic Fatigue Syndrome. An Open-Label Phase II Study with Rituximab Maintenance Treatment. PLoS One. 2015 Jul 1;10(7):e0129898. doi: 10.1371/journal.pone.0129898. eCollection 2015. PMID 26132314